CLINICAL TRIAL: NCT03539549
Title: Evaluation of Abicipar Pegol in Patients With Neovascular Age-related Macular Degeneration
Brief Title: A Study to Evaluate Abicipar Pegol for Safety and Treatment Effect in Participants With Neovascular Age-related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1771-201-008
Record Dates: First submitted 2018-05-17; First posted 2018-05-29 (Actual); Results first posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — abicipar pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Abicipar pegol 2 mg (Experimental): Abicipar pegol 2 mg administered to the study eye by intravitreal injection on Day 1 and Weeks 4, 8, 16, and 24.
  Interventions: Drug: Abicipar pegol

INTERVENTIONS:
Drug: Abicipar pegol — Abicipar pegol 2 mg administered to the study eye by intravitreal injection on Day 1 and Weeks 4, 8, 16, and 24.

SUMMARY:
The objective of this study is to evaluate abicipar pegol for safety and treatment effects in participants with neovascular age-related macular degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, 50 years of age or older at the time of informed consent
* Best Corrected Visual Acuity (BCVA) ≤ 78 and ≥ 24 letters (20/32 to 20/320 Snellen equivalents, respectively) at Screening and at Baseline (Day 1, prior to treatment) visits in the study eye
* BCVA of 34 letters (Snellen equivalent 20/200) or better at Baseline (Day 1, prior to treatment) in the non-study eye

Exclusion Criteria:

* Active periocular, ocular, or intraocular infection at baseline (Day 1) (either eye)
* Previous or concurrent macular laser treatment (study eye)
* Cataract or refractive surgery within 3 months prior to baseline (study eye)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Li, MD, Study Director — Allergan
Locations (37):
- United States (37):
  - Barnet Dulaney Perkins Eye Center, Phoenix, Arizona
  - Retina Associates Southwest, PC, Tucson, Arizona
  - Win Retina, Arcadia, California
  - Retina Consultants of Orange County, Fullerton, California
  - Mark B. Kislinger, MD, Inc., Glendora, California
  - Atlantis Retina Institute (Atlantis Eyecare), Huntington Beach, California
  - N. California Retina Vitreous Associates Medical Group, INC., Mountain View, California
  - California Eye Specialists Medical Group, Inc, Pasadena, California
  - Retinal Consultants Medical Group, Inc., Sacramento, California
  - Colorado Retina Associates, Golden, Colorado
  - Retina Specialty Institute, Pensacola, Florida
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Georgia Retina, P.C., Marietta, Georgia
  - Marietta Eye Clinic, Marietta, Georgia
  - Gailey Eye Clinic, Bloomington, Illinois
  - Raj K. Maturi, MD, PC, Indianapolis, Indiana
  - Sabates Eye Center, Leawood, Kansas
  - Sierra Eye Associates, Reno, Nevada
  - Capital Region Retina, PLLC, Albany, New York
  - Ophthalmic Consultants of Long Island, Lynbrook, New York
  - Retina Associates of Western New York, Rochester, New York
  - Retina Vitreous Surgeons of Central NY, P.C., Syracuse, New York
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Pennsylvania Retina Specialists, P.C., Camp Hill, Pennsylvania
  - Charleston Neuroscience Institute, Ladson, South Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Retina Research Institute of Texas, Abilene, Texas
  - Texas Retina Associates, Arlington, Texas
  - Austin Retina Associates, Austin, Texas
  - Texan Eye, Austin, Texas
  - Retinal Consultants of Houston, Houston, Texas
  - Premiere Retina Specialists, Midland, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas
  - Retina Consultants of Houston, The Woodlands, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
  - Retina Institute of Virginia, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 124 participants were enrolled in the study. Out of 124, one participant was not treated with study drug and was subsequently discontinued from the study. The participant was not included in the Safety Population or analyses.
Period: Overall Study
Arm/Group | Abicipar Pegol 2 mg
Started | 123
Completed | 106
Not Completed | 17
Not completed — Adverse Event | 12
Not completed — Lost to Follow-up | 1
Not completed — Death | 2
Not completed — Progressive Disease | 1
Not completed — Reason not Specified | 1

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received at least 1 administration of study treatment.
Arm/Group | Abicipar Pegol 2 mg
Number analyzed (Participants) | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.3 (8.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 119
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 119
  More than one race | 0
  Unknown or Not Reported | 0
Best Corrected Visual Acuity (BCVA) [Mean (Standard Deviation); unit: letters] — BCVA was measured using an eye chart and reported as number of letters read correctly using Early Treatment of Diabetic Retinopathy Study (ETDRS) Scale (ranging from 0 to 100 letters) in study eye. Lower number of letters read correctly on eye chart, worse the vision (or visual acuity). Study eye: eye that meets entry criteria. If both eyes met entry criteria, eye with worse BCVA at baseline (Day 1) was selected as study eye. If both eyes had same BCVA values at baseline (Day 1), then participant had to select their non-dominant eye for treatment, or else right eye was selected. Population: Number analyzed is the number of participants with BCVA data available at baseline.
  letters
    number analyzed (Participants) | 122
    (all) | 62.0 (12.19)
Central Retinal Thickness (CRT) [Mean (Standard Deviation); unit: microns] — CRT was assessed using spectral domain optical coherence tomography (SD-OCT), a non-invasive diagnostic system providing high-resolution imaging sections of the retina. SD-OCT was performed in the study eye after pupil dilation. The study eye is defined as the eye that meets the entry criteria. If both eyes met the entry criteria, the eye with the worse BCVA at baseline (Day 1) was selected as the study eye. If both eyes had same BCVA values at baseline (Day 1), then the participant had to select their non-dominant eye for treatment, or else the right eye was selected as the study eye. Population: Number analyzed is the number of participants with CRT data available at Baseline.
  microns
    number analyzed (Participants) | 122
    (all) | 353.1 (94.05)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Stable Vision
Description: Stable vision was defined as a loss of fewer than 15 letters in Best Corrected Visual Acuity (BCVA) compared to baseline. BCVA was measured using an eye chart and is reported as the number of letters read correctly using the Early Treatment of Diabetic Retinopathy Study (ETDRS) Scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved. The study eye was defined as the eye that meets the entry criteria. If both eyes met the entry criteria, the eye with the worse BCVA at baseline (Day 1) was selected as the study eye. If both eyes had same BCVA values at baseline (Day 1), then the participant had to select their non-dominant eye for treatment, or else the right eye was selected as the study eye.
Time Frame: Baseline (Day 1) to Week 28
Population: Safety Population included all participants who received at least 1 administration of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abicipar Pegol 2 mg
Number analyzed (Participants) | 123
percentage of participants | 97.6 [94.2 to 99.8]

2. Secondary Outcome: Change From Baseline in Central Retinal Thickness (CRT) in the Study Eye
Description: CRT was assessed using spectral domain optical coherence tomography (SD-OCT), a non-invasive diagnostic system providing high-resolution imaging sections of the retina. SD-OCT was performed in the study eye after pupil dilation. A negative change from Baseline indicated improvement. The study eye is defined as the eye that meets the entry criteria. If both eyes met the entry criteria, the eye with the worse BCVA at baseline (Day 1) was selected as the study eye. If both eyes had same BCVA values at baseline (Day 1), then the participant had to select their non-dominant eye for treatment, or else the right eye was selected as the study eye.
Time Frame: Baseline (Day 1) to Week 28
Population: Safety Population included all participants who received at least 1 administration of study treatment. Number analyzed is the number of participants with data available at the given time point.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Abicipar Pegol 2 mg
Number analyzed (Participants) | 123
microns | -82.5 (102.13)

3. Secondary Outcome: Percentage of Participants With Loss of 15 or Less EDTRS Letters in BCVA From Baseline in the Study Eye
Description: BCVA was measured using an eye chart and is reported as the number of letters read correctly using the ETDRS Scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved. The study eye was defined as the eye that meets the entry criteria. If both eyes met the entry criteria, the eye with the worse BCVA at baseline (Day 1) was selected as the study eye. If both eyes had same BCVA values at baseline (Day 1), then the participant had to select their non-dominant eye for treatment, or else the right eye was selected as the study eye.
Time Frame: Baseline (Day 1) to Week 28
Population: Safety Population included all participants who received at least 1 administration of study treatment. Overall number of participants analyzed are the participants with data available for analyses.
Measure: Number; unit: percentage of participants
Arm/Group | Abicipar Pegol 2 mg
Number analyzed (Participants) | 106
percentage of participants | 0.9

4. Secondary Outcome: Change Form Baseline in BCVA in the Study Eye
Description: as for outcome 3
Time Frame: Baseline (Day 1) to Week 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Abicipar Pegol 2 mg
Number analyzed (Participants) | 106
letters | 3.6 (7.19)

5. Secondary Outcome: Percentage of Participants With a Gain of 15 or More ETDRS Letters in BCVA From Baseline in the Study Eye
Description: as for outcome 3
Time Frame: Baseline (Day 1), Week 28
Population: Safety Population included all participants who received at least 1 administration of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abicipar Pegol 2 mg
Number analyzed (Participants) | 123
percentage of participants | 9.8 [5.2 to 16.6]

6. Other Pre Specified Outcome: Percentage of Participants With Change From Baseline in Full Ophthalmic Exam Findings [i.e. Slit Lamp Exam, Intraocular Pressure (IOP) Measurements, Funduscopic Exam]
Time Frame: Baseline to Week 28
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Changes From Baseline in General Physical Condition as Measured Through General Physical Exam
Time Frame: Baseline to Week 28
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Percentage of Participants With Changes From Baseline in Vital Signs (Blood Pressure, Pulse Rate, ECG)
Time Frame: Baseline to Week 28
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Percentage of Participants With Change From Baseline in Clinically Relevant Laboratory Values (Serum Chemistry, Hematology, Urinalysis)
Time Frame: Baseline to Week 28
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Percentage of Participants With Anti-abicipar Antibodies Measured in Serum
Time Frame: Baseline to Week 28
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From first dose up to 28 weeks
Description: Safety Population included all participants who received at least 1 administration of study treatment.
Arm/Group | Abicipar Pegol 2 mg
All-Cause Mortality (participants affected / at risk) | 2/123
Serious Adverse Events (participants affected / at risk) | 16/123
Other Adverse Events (participants affected / at risk) | 0/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abicipar Pegol 2 mg (N=123)
Atrial fibrillation (Cardiac disorders) | 2
Tachyarrhythmia (Cardiac disorders) | 1
Iritis (Eye disorders) | 1
Retinal haemorrhage (Eye disorders) | 1
Vitreous haemorrhage (Eye disorders) | 1
Vitritis (Eye disorders) | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2018-10-16): https://cdn.clinicaltrials.gov/large-docs/49/NCT03539549/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/49/NCT03539549/SAP_001.pdf